CLINICAL TRIAL: NCT07348172
Title: Characterizing Drug Liking During Drug Administration in Peri-procedural Clinical Settings
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Patrick Purdon, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB-80824
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Drug Liking
MeSH Terms: interventions — Amisulpride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug (Experimental): Participants receive study drug prior to fentanyl administration before their procedure.
  Interventions: Drug: Amisulpride
- Placebo (Placebo Comparator): Participants receive placebo prior to fentanyl administration before their procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amisulpride — Medication administered as a single intravenous dose.
  Arms: Drug
Drug: Placebo — Matching Placebo given by single intravenous (IV) administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether medications used in peri-procedural clinical settings can modulate drug liking.

DETAILED DESCRIPTION:
Specifically, we aim to measure differences in drug liking with a VAS (0 - 100) questionnaire. Additionally, we will monitor neural activity recording a frontal electroencephalogram (EEG) to detect changes in brain signals associated with opioid drug effects. By comparing behavioral and neurophysiological data across treatment and control groups, this study seeks to explore the therapeutic potential of this medication.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification of I, II or III
* Candidates who are expected to receive fentanyl up to 3 mcg/kg IBW for their scheduled for surgery or procedure

Exclusion Criteria:

* Craniofacial abnormalities
* Known or suspected difficult intubation or mask ventilation
* Known or suspected need for rapid sequence induction and intubation
* Allergies or hypersensitivities to amisulpride or fentanyl
* Clinically significant pulmonary disease, such as chronic obstructive lung disease requiring long-term oxygen therapy, or other conditions that, in the study team's judgment, may increase the risk of severe respiratory depression with opioid administration
* History of long QT syndrome
* Any heart rhythm other than normal sinus rhythm (including but not limited to atrial fibrillation, atrial flutter, paced rhythms, ventricular tachycardia, or any supraventricular tachycardia)
* History of Torsades de Pointes
* History of psychosis
* History of movement disorders e.g. Parkinson's Disease
* Past chronic use of anti-psychotics
* Current use of amisulpride, droperidol, levodopa, lithium, clozapine, metoclopramide, benzodiazepines
* Current use of opioids
* History of opiate abuse within the last 3 years
* Known or suspected severe chronic pain condition that require use of opiates or limit daily activities
* History of pheochromocytoma
* History of concomitant prolactin-dependent tumors e.g. prolactinoma, breast cancer
* Pregnancy or nursing
* Failure to satisfy the investigator of fitness to participate for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Drug Liking Rating | One minute before and 1, 3, and 5 minutes after fentanyl administration
  Change in drug liking rating (0-100), anchored by divert "not at all=0" and "as much as possible=100".

SECONDARY OUTCOMES:
EEG band power | From administration of the study drug to about 1 hour after.
  Assessment of the change in power of the frontal EEG canonical frequency bands measured in decibles (dB).
Change in Sedation Rating | One minute before and 1, 3, and 5 minutes after fentanyl administration
  Change in self-reported sedation rating (0-100), anchored by divert "not at all=0" and "as much as possible=100".

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No